CLINICAL TRIAL: NCT06863181
Title: Comparison of the Effectiveness of Conventional and Cooled Radiofrequency Ablation in Advanced Knee Osteoarthritis
Brief Title: Comparison of Conventional and Cooled Radiofrequency Ablation in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Naz Kalem, specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-064
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Radiofrequency Ablation (Active Comparator): Conventional radiofrequency ablation with fluoroscopy
  Interventions: Device: Radiofrequency ablation
- Cooled Radiofrequency Ablation (Experimental): Cooled radiofrequency ablation with ultrasound
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — Genicular nerve neurolysis with heat

SUMMARY:
The aim of this study was to examine and compare the effects of conventional and cooled radiofrequency ablation on pain and disability levels in patients with knee pain resistant to other treatments due to knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain lasting more than 6 months
* Age between 50 and 80
* Diagnosis of radiographically proven grade III or IV knee osteoarthritis according to the Kellgren-Lawrence Grading Scale, marked narrowing of the medial compartment of the tibiofemoral joint space
* Presence of pain resistant to conservative treatment

  * Exercise
  * Physical therapy agents
  * Use of oral anti-inflammatory agents

Exclusion Criteria:

* History of trauma to the knee area
* History of knee surgery
* Presence of systemic inflammatory disease affecting the knee joint
* Presence of peripheral neuropathy or radiculopathy
* Pregnancy
* Hemodynamic instability
* Presence of skin or soft tissue infection at the injection site
* Refusal to participate in the study
* Presence of acute knee pain with accompanying inflammatory findings
* Presence of a serious psychiatric disorder or neurological disease Having received an intra-articular injection within the last 3 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before treatment (0. week), 4 weeks after treatment (4.week), 12 weeks after treatment (12.week)
  Patients will select their pain from 10 mm scale

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Before treatment (0. week), 4 weeks after treatment (4.week), 12 weeks after treatment (12.week)
  This scale about patient's disability due to knee osteoarthritis
5-Point Likert Patient Satisfaction Scale | Before treatment (0. week), 4 weeks after treatment (4.week), 12 weeks after treatment (12.week)
  '0' =I am not happy at all, '5'=I am very pleased
Change in frequency of analgesic use | Before treatment (0. week), 4 weeks after treatment (4.week), 12 weeks after treatment (12.week)
  How many analgesic did use in past week?

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)